CLINICAL TRIAL: NCT00991133
Title: A Phase 1, Open-Label, Multi-Center Safety and Tolerability Pilot Combination Study of Clofarabine, Etoposide, Cyclophosphamide, PEG-asparaginase, and Vincristine in Pediatric Patients With Acute Lymphoblastic Leukemia (ALL) in First Relapse
Brief Title: A Safety and Tolerability Study of Clofarabine, Etoposide, Cyclophosphamide, PEG-asparaginase, and Vincristine in Pediatric Acute Lymphoblastic Leukemia (ALL)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLO08808
Record Dates: First submitted 2009-10-05; First posted 2009-10-07 (Estimated); Last update posted 2015-04-30 (Estimated); Status verified 2015-04

CONDITIONS: Lymphoblastic Leukemia, Acute, Childhood
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Clofarabine; Etoposide; Cyclophosphamide; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Clofarabine (Experimental): Patients received a maximum of 2 cycles of the intravenous (IV) 5-drug regimen (clofarabine, etoposide,cyclophosphamide, PEG-asparaginase, and vincristine) plus intrathecal methotrexate, and then entered follow-up. Patients who achieved complete remission (CR) or complete remission with incomplete platelet recovery (CRp) after 1 cycle of study drugs were eligible to receive a second cycle of study drugs upon recovery of peripheral blood counts, and patients who did not have leukemic progression were eligible to receive a second treatment cycle at the investigator's discretion.
  Interventions: Drug: Clofarabine incorporated into a 5-drug regimen

INTERVENTIONS:
Drug: Clofarabine incorporated into a 5-drug regimen — Clofarabine (IV) 40mg/m2 into an intensive chemotherapy regimen of etoposide, cyclophosphamide, PEG-asparaginas, and vincristine
  Other Names: Clolar; VP-16; Cytoxan; PEGaspar-aginase; Oncovin

SUMMARY:
This is an open-label study of Clofarabine, Etoposide, Cyclophosphamide, PEG-asparaginase, and Vincristine to assess this 5-drug treatment's safety and tolerability in pediatric patients with first relapse Acute Lymphoblastic Leukemia (ALL).

DETAILED DESCRIPTION:
The trial is a Phase 1, open-label study to assess the safety and tolerability of incorporating clofarabine into an intensive chemotherapy regimen of etoposide, cyclophosphamide, PEG-asparaginase, and vincristine. Patients enrolled in this study will receive a maximum of 2 cycles of the 5-drug regimen, then will be treated according to investigator discretion. After the study treatment period, all patients will be followed for a minimum of 4 months beyond the final study visit. This study will include a maximum of 12 evaluable patients.

ELIGIBILITY:
Inclusion Criteria:

* Be in first relapse with >25% blasts in the bone marrow with a duration of first remission of ≥6 months and no longer in the intensive phase(s) of initial ALL therapy (e.g., patients who are in the maintenance or continuation phases of therapy [or beyond] and who have completed the induction or intensification phases).
* Have received no more than 2 prior induction regimens prior to the date of first relapse. Patients who are in first relapse but have failed a re-induction attempt (i.e., 1 cycle of re-induction therapy) are not eligible for inclusion in this study.
* Be ≥1 and ≤30 years old and have a body weight of >10 kg at study entry. (Note: no more than 3 patients aged >21 ≤30 are to be enrolled.)
* Be able to receive all study drugs with no known contra-indications.
* Be able to provide adequate venous access.
* Have a Karnofsky Performance Status (KPS) of ≥50 for patients >10 years of age or a Lansky Performance Status (LPS) of ≥50 for patients ≤10 years of age.
* Patients (≥18 years of age) or the parent or legal guardian(s) (for patients <18 years of age) must provide signed, written informed consent according to local institutional review board (IRB) and institutional requirements. For patients <18 years of age, signed assent should be obtained according to local IRB and institutional requirements.
* Be able to comply with study procedures and follow-up examinations.
* Have adequate liver, renal, pancreatic, and cardiac function considered acceptable by laboratory values and cardiac assessments
* Have no active central nervous system (CNS) leukemia, as evidenced by negative cytology on lumbar puncture and absence of clinical central neurologic symptoms. Diagnostic lumbar puncture should be performed only after all other eligibility assessments have been completed and reviewed, except for bone marrow aspirate and/or biopsy. Patients with CNS1 or CNS2 leukemia may be enrolled in the study.
* Have recovered to baseline from all toxicities from prior chemotherapy regimens prior to enrollment in the study.

Exclusion Criteria:

* Have received previous treatment with clofarabine.
* Have a history of clinical allergy (Grade 3 or 4) to PEG-asparaginase.
* Have a history of severe pancreatitis (Grade 3 or 4) attributed to asparaginase therapy.
* Have Burkitt's leukemia.
* Have overt testicular relapse.
* Adequate time has not elapsed since patient's last therapy. Patients who relapse while receiving standard ALL maintenance chemotherapy will not be required to have a washout period before entry onto this study. Note that patients may receive intrathecal (IT) ara-C, methotrexate, or hydrocortisone immediately prior to the administration of study drugs. Patients may also receive hydroxyurea up to 24 hours prior to the start of study therapy. Patients who relapse when they are not receiving standard ALL maintenance therapy must have fully recovered from the acute toxic effects of all prior therapy (excluding hematologic toxicity), immunotherapy or radiotherapy.
* Have an uncontrolled systemic fungal, bacterial, viral, or other infection. For patients with a history of fever within the preceding 3 days at the time of enrollment, documentation of negative blood cultures for at least 48 hours is required.
* Are pregnant or lactating.
* Male and female patients who are fertile must agree to use an effective means of birth control (i.e., latex condom, diaphragm, cervical cap, etc.) while on study therapy, and for a minimum of 1 month following final study visit.
* Have psychiatric disorders that would interfere with consent, study participation, or follow-up.
* Have any other severe concurrent disease, or have a history of serious organ dysfunction or disease involving the heart, kidney, liver, or pancreas.
* Have received any stem cell transplantation or high-dose chemotherapy with stem cell rescue regimen.
* Have a history of cirrhosis or known human immunodeficiency virus (HIV)/acquired immunodeficiency syndrome (AIDS).
* Have a history of at least 1 positive test for hepatitis B or hepatitis C infection.
* Have Down syndrome.
* Are currently participating in another concurrent investigational treatment protocol.

Ages: 1 Year to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 8 (Actual)
Dates: Start 2009-10; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
The incidence of DLTs (Dose Limiting Toxicities) experienced with 1 cycle of this 5-drug regimen in this patient population (in all patients who receive any doses of study drugs) | 1 cycle

SECONDARY OUTCOMES:
Overall toxicity profile documented by incidence of AEs, SAEs, and/or DLTs | 1 cycle
Efficacy as documented by complete remission (CR), time and duration of remission, event-free survival (EFS), 4-month EFS, disease-free survival (DFS), and overall survival | 2 cycles

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (6):
- United States (6):
  - Children's Hospital Los Angeles, Los Angeles, California
  - The Children's Hospital, Aurora, Colorado
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Children's Memorial Hospital, Chicago, Illinois
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Seattle Children's Hospital, Seattle, Washington